CLINICAL TRIAL: NCT00002627
Title: PHASE I/II TRIAL OF THE ADDITION OF TAXOL TO HIGH DOSE CARBOPLATIN AND CYCLOPHOSPHAMIDE WITH AUTOLOGOUS PERIPHERAL BLOOD PROGENITOR CELL SUPPORT IN PATIENTS WITH HIGH RISK STAGE II AND III BREAST CANCER
Brief Title: Addition of Paclitaxel to High-Dose Combination Chemotherapy in Treating Patients With High-Risk Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Louis University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064016; SLUMC-8038; NCI-V95-0607
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2000-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Mesna; Paclitaxel; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: mesna
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells, allowing higher doses of chemotherapy to be used.

PURPOSE: Phase I/II trial to study the effectiveness of paclitaxel when added to high-dose combination chemotherapy followed by peripheral stem cell transplantation in treating women with breast cancer at high risk of relapse.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose of paclitaxel when given with high-dose carboplatin/cyclophosphamide with autologous peripheral blood stem cell support in women with high-risk stage II/III breast cancer. II. Assess the nonhematologic toxicities associated with this combination. III. Assess the progression-free and overall survival of these patients following this treatment.

OUTLINE: This is a dose-finding study. All patients undergo collection of peripheral blood stem cells (PBSC) with granulocyte colony-stimulating factor (G-CSF) mobilization prior to high-dose chemotherapy. Cohorts of 3-5 patients are treated at successively higher dose levels of paclitaxel until a maximum tolerated dose (MTD) is found. Paclitaxel is given as a single 6-hour infusion, followed by fixed doses of high-dose cyclophosphamide for 2 days, then carboplatin for 3 days. Four days later, patients receive PBSC and G-CSF for hematopoietic reconstitution. Additional patients are entered at the MTD. Patients are followed every 3 months for 1 year, every 4 months for 1 year, then every 4-6 months thereafter.

PROJECTED ACCRUAL: It is expected that 24-30 patients will be accrued; a study duration of 1-1.5 years is anticipated.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed adenocarcinoma of the breast of the following stages: Stage II/IIIA disease with 4 or more involved axillary lymph nodes Stage IIIB Inflammatory No bone marrow involvement documented on bone marrow aspiration and biopsy Prior breast cancer allowed Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 65 Sex: Women only Menopausal status: Not specified Performance status: Karnofsky 70%-100% Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine clearance at least 60 mL/min Cardiovascular: Left ventricular ejection fraction at least 50% by MUGA No abnormal cardiac conduction documented as second- or third-degree heart block or bundle branch block Pulmonary: DLCO at least 60% of predicted Other: Not HIV positive No history of second malignancy within 5 years except: Nonmelanomatous skin cancer In situ carcinoma of the cervix No pregnant women

PRIOR CONCURRENT THERAPY: At least 3 courses of induction therapy required, with regimen at the discretion of the investigator No disease progression during induction

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1994-11

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Petruska, MD, Study Chair — St. Louis University
Locations (1):
- St. Louis University Health Sciences Center, St Louis, Missouri, United States